CLINICAL TRIAL: NCT02399657
Title: A Single Arm, Single Dose Study to Evaluate the Effect of Intravitreal Dexamethasone Implant (Ozurdex®) on Hard Exudates of Diabetic Macular Edema
Brief Title: Effect of Dexamethasone Implant in Hard Exudate Complicated With Diabetic Macular Edema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Hyun Woong Kim, Associate professor, Inje University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXTINCT
Record Dates: First submitted 2015-03-18; First posted 2015-03-26 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus; Macular Edema; Retinal Exudates and Deposits
Keywords: diabetes mellitus; macular edema; hard exudate; intravitreal injections; dexamethasone; implant
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Drug Implants; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravitreal dexamethasone implant (Experimental): Intravitreal dexamethasone 0.7mg implant (Ozurdex)
  Interventions: Drug: Intravitreal dexamethasone 0.7mg implant

INTERVENTIONS:
Drug: Intravitreal dexamethasone 0.7mg implant — Ozurdex at day 0 (fixed), 5 months (fixed), 10 months pro re nata or 11 months pro re nata
  Other Names: Ozurdex injection

SUMMARY:
A Single Arm, Single Dose Study to Evaluate the Effect of intravitreal dexamethasone implant (Ozurdex®) on hard exudates of diabetic macular edema.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) is important vision threatening complication of diabetes mellitus. Laser photocoagulation, vitrectomy, intravitreal steroid injection and intravitreal antiVEGF (anti vascular endothelial growth factor) injection are being used as treatment of DME. Sustained releasing intravitreal dexamethasone implant has been known to be effective in reducing the central retinal thickness and gain of vision for DME. Although hard exudate at macula is important pathology of DME, impact of intravitreal dexamethasone implant on hard exudate are not studied yet. Therefore the investigators designed the descriptive study to reveal the hard exudate change in DME eyes treated with intravitreal dexamethasone implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with CSME (clinically significant macular edema) with hard exudates within 1500 micrometer from foveal center
2. Those who have a BCVA (best corrected visual acuity) of study eye between 0.06(20/320) and 0.5(20/40)
3. Those who have a central macular thickness on OCT over 300 micrometer
4. If both eyes are eligible, eye having more hard exudates is selected (contralateral eye should be treated with corticosteroid other than Ozurdex or focal laser photocoagulation, anti-VEGF (vascular endothelial growth factor) injection is not allowed in contralateral eye)

Exclusion Criteria:

1. Those who have CSME without hard exudates
2. Those who have macular edema not related with diabetic retinopathy (e.g. AMD (age-related macular degeneration), uveitis, retinal vein occlusion and untreated malignant hypertension)
3. Those who have a history of Intraocular surgery (e.g. cataract surgery) within 3 months
4. Those who have a visual acuity of contralateral eye less than 0.1 (10/100)
5. Those who received focal laser treatment on macula within 3 months
6. Those who had intravitreal anti-VEGF agent injection within 3 months
7. Those who had intravitreal triamcinolone injection within 6 months
8. Those who have other ophthalmologic disease affecting visual acuity (e.g. central corneal opacity, cataract change at lens center)
9. Those who have severe systemic disease (e.g. uncontrolled DM, hypertension, cardiovascular disease, cerebrovascular disease)
10. Those who refuse to submit written consent
11. Those who cannot understand the contents of the clinical study and cooperate in the clinical trial
12. Those who are pregnant or lactating women
13. Those who have a history of vitrectomy
14. Those who require systemic corticosteroid or immunosuppressive agent treatment
15. Those who are banned from using Ozurdex

    * Ocular infection or periocular infection
    * Advanced glaucoma
    * Hypersensitivity to dexamethasone or other component of Ozurdex
    * Posterior lens capsule rupture or Aphakia
    * Anterior chamber intraocular lens or posterior capsule rupture

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The ratio of eyes showing reduced hard exudates in macula (1500 micrometer from foveal center) | after 12 months

SECONDARY OUTCOMES:
The average change in ETDRS (Early Treatment Diabetic Retinopathy Study) visual acuity | after 12 months
The Ratio of eyes with central macular thickness under 290 micrometer in OCT (optical coherence tomography) | after 12 months
The Ratio of eyes showing reduced perifoveal capillary leakage in fluorescein angiography | after 12 months
The average change in number of microaneurysm in macula | after 12 months
The progression rate of cataract | for 12 months
Number of eyes having increased intraocular pressure | for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Woong Kim, M.D., Study Director — Inje University; Ji Eun Lee, M.D., Principal Investigator — Pusan National University Hospital; Joo Eun Lee, M.D., Principal Investigator — Inje University Haeundae Paik Hospital; Woo Jin Jeung, M.D., Principal Investigator — Dong-A University Hospital; Sang Joon Lee, M.D., Principal Investigator — Kosin University Gospel Hospital; In Young Chung, M.D., Principal Investigator — Gyeongsang National University Hospital; Jae Pil Shin, M.D., Principal Investigator — Kyungpook National University Hospital; Woo Hyok Chang, M.D., Principal Investigator — Yeungnam University Hospital
Locations (8):
- South Korea (8):
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Kosin University Gospel Hospital, Busan
  - Dong-A University hospital, Busan
  - Pusan national university hospital, Busan
  - Inje University Haeundae Paik hospital, Busan
  - Inje University Busan Paik hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu

REFERENCES:
- [Background] Bhagat N, Grigorian RA, Tutela A, Zarbin MA. Diabetic macular edema: pathogenesis and treatment. Surv Ophthalmol. 2009 Jan-Feb;54(1):1-32. doi: 10.1016/j.survophthal.2008.10.001. PMID 19171208
- [Background] Klein R, Klein BE, Moss SE, Cruickshanks KJ. The Wisconsin Epidemiologic Study of Diabetic Retinopathy. XV. The long-term incidence of macular edema. Ophthalmology. 1995 Jan;102(1):7-16. doi: 10.1016/s0161-6420(95)31052-4. PMID 7831044
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Haller JA, Kuppermann BD, Blumenkranz MS, Williams GA, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Randomized controlled trial of an intravitreous dexamethasone drug delivery system in patients with diabetic macular edema. Arch Ophthalmol. 2010 Mar;128(3):289-96. doi: 10.1001/archophthalmol.2010.21. PMID 20212197
- [Derived] Yoon CK, Sagong M, Shin JP, Lee SJ, Lee JE, Lee JE, Chung I, Jeong WJ, Pak KY, Kim HW. Title: efficacy of intravitreal dexamethasone implant on hard exudate in diabetic macular edema. BMC Ophthalmol. 2021 Jan 15;21(1):41. doi: 10.1186/s12886-020-01786-2. PMID 33451297